CLINICAL TRIAL: NCT01550393
Title: Discovery and Validation of Wilms Tumor Markers Using Urine Proteomics
Brief Title: Biomarkers in Urine Samples From Patients With Wilms Tumor
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: AREN12B4; COG-AREN12B4 (Other: Children's Oncology Group); CDR0000727337 (Other: Clinical Trials.gov); AREN12B4 (Other: Children's Oncology Group); NCI-2012-00702 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2012-03-06; First posted 2012-03-12 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-07

CONDITIONS: Kidney Cancer
Keywords: stage II Wilms tumor; stage III Wilms tumor; recurrent Wilms tumor and other childhood kidney tumors
MeSH Terms: conditions — Kidney Neoplasms; Wilms Tumor | interventions — Enzyme-Linked Immunosorbent Assay

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Urine
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: proteomic profiling
Other: enzyme-linked immunosorbent assay
Other: laboratory biomarker analysis
Other: medical chart review

SUMMARY:
RATIONALE: Studying samples of urine from patients with cancer in the laboratory may help doctors identify biomarkers related to cancer.

PURPOSE: This clinical trial studies biomarkers in urine from patients with Wilms tumor.

DETAILED DESCRIPTION:
OBJECTIVES:

* To validate the prognostic performance of specific-candidate Wilms tumor markers by measuring their urinary concentration using enzyme-linked immunosorbent assays (ELISAs) in urine specimens collected at diagnosis from 50 patients with favorable histology Wilms tumor who relapsed and 50 patients who did not relapse.

OUTLINE: Urine specimens are analyzed using enzyme-linked immunosorbent assays (ELISAs) for biomarkers.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Urine specimens collected at diagnosis will be selected from patients with stage II-III Wilms tumors, with both local and non-local sites of disease relapse
* Clinical patient information (urinalysis/macro, age, gender, congenital defects/syndromes, comorbidities, tumor stage, size, pathology, therapy, outcome) available

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Max Age: 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with stage II-III Wilms tumors
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2012-03; Primary Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Wilms tumor biomarkers identified by ELISA

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth A. Mullen, MD, Principal Investigator — Dana-Farber Cancer Institute